CLINICAL TRIAL: NCT03990714
Title: Intracorporeal Vs Extracorporeal Anastomosis in Patients Undergoing Laparoscopic Right Hemicolectomy: a Multicenter Randomized Clinical Trial (The IVEA-study)
Brief Title: Intracorporeal Vs Extracorporeal Anastomosis in Laparoscopic Right Hemicolectomy
Acronym: IVEA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Torrecárdenas (Other)
Collaborators: Sponsor- Investigator MD Ángel Reina Duarte. HUTorrecárdenas (Unknown); Sponsor-Investigator BA Francisco Rubio Gil. HU Torrecárdenas (Unknown); Sponsor-Investigator MD Elisabet Vidaña Márquez. HU Torrecárdenas (Unknown); Sponsor-Investigator MD Juan Manuel García Torrecillas. HU Torrecárdenas (Unknown); Sponsor-Investigator Rocío Torres Fernández. HU Torrecárdenas (Unknown); Sponsor-Investigator MD Almudena Moreno Serrano. Hospital Inmaculada. Huercal-Overa (Unknown); Sponsor-Investigator MD Pedro Moya Forcén. HU Torrecárdenas (Unknown); Sponsor-Investigator MD Jorge Alejandro Benavides Buleje. HU Reina Sofía (Unknown)
Responsible Party: Principal Investigator, Manuel Ferrer Márquez, MD, Hospital Universitario Torrecárdenas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUTorrecardenas
Record Dates: First submitted 2019-06-12; First posted 2019-06-19 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Colorectal Surgery; Anastomotic Leak; Colectomy; Laparoscopy
Keywords: Right hemicolectomy; Intracorporeal anastomosis; Extracorporeal anastomosis; Laparoscopy
MeSH Terms: conditions — Anastomotic Leak

STUDY DESIGN:
Intervention Model Description: The IVEA-study is a prospective multicenter randomized trial with two parallel groups being done IA or EA in laparoscopic right hemicolectomy for right colon neoplasia.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intracorporeal anastomosis (Experimental): The specimen was preferentially extracted via a small Pfannenstiel-type incision with the protection of an Alexis Wound Protector (Applied Medical, Rancho Santa Margarita, California, USA). The incision for the extraction of the right colon is sutured in two layers by absorbable suture. The ileum was held by the assistant to prevent rotation of its mesentery. A stay suture was applied 10 cm proximal and distal to the stapled ends of the terminal ileum and colon, respectively, and then held by the assistant. An enterotomy and colotomy were made sharply at the antimesenteric corner of the staple lines. An isoperistaltic side-to-side anastomosis was fashioned with a 60-mm laparoscopic stapler. A 2-0 double-barbed suture was used to close the enterocolotomy, in two planes (the first submucosal, and the second sero-serous). The mesenteric defect and the mesocolon after the construction of either type of anastomosis were not closed. Drains were not used routinely.
  Interventions: Procedure: Right hemicolectomy
- Extracorporeal anastomosis (Experimental): The mobilized colon was externalized preferentially via a transverse or midline incision with the protection of an Alexis Wound Protector (Applied Medical, Rancho Santa Margarita, California, USA). A stay suture was applied 10 cm proximal and distal to the stapled ends of the terminal ileum and colon. An enterotomy and colotomy were made sharply at the antimesenteric corner of the staple lines. An isoperistaltic side-to-side anastomosis was fashioned with a 60-mm laparoscopic stapler. A 2-0 double-barbed suture was used to close the enterocolotomy, in two planes (the first submucosal, and the second sero-serous). The mesenteric defect and the mesocolon after the construction of either type of anastomosis were not closed.The incision for the extraction of the right colon and the realization of the anastomosis is sutured in two layers by absorbable suture. Drains were not used routinely.
  Interventions: Procedure: Right hemicolectomy

INTERVENTIONS:
Procedure: Right hemicolectomy — It is the resection of the right colon by a tumor and the reconstruction by an ileocolic anastomosis: intracorporeal or extracorporeal

SUMMARY:
Objective. The aim of this study was to evaluate short-term outcomes of performing intracorporeal versus extracorporeal anastomosis in laparoscopic right hemicolectomy for right colon neoplasm. Background. Despite advances in laparoscopic approach in colorectal surgery and the clear benefit of this approach over open surgery, the technical difficulty in performing intracorporeal anastomosis causes certain groups continue performing it extracorporeally in right colon surgery.

Methods. This study was a prospective multicenter randomized trial with two parallel groups being done intracorporeal anastomosis (IA) or extracorporeal anastomosis (EA) in laparoscopic right hemicolectomy for right colon neoplasm, carried out between January 2016 and December 2018.

DETAILED DESCRIPTION:
Right hemicolectomy using a minimally invasive technique allows for an earlier recovery, with less postoperative pain and less hospital stay. After right hemicolectomy, the ileocolic anastomosis is not performed "naturally" as is habitually done in low anterior resections or sigmoidectomies. There is, therefore, no standardization in the reconstruction technique, with two possibilities: intracorporeal and extracorporeal anastomosis.

The intracorporeal anastomosis allows proper visualization of it, ensuring adequate conformation (absence of rotation or traction), in addition allowing the closure of the mesos and avoiding the possible appearance of internal hernia, also allowing to choose the location and length of the incision necessary for the extraction of the piece. On the other hand, it is a difficult technique that requires high training in advanced laparoscopy.

The extracorporeal anastomosis is performed by extracting both ends (terminal ileum and transverse colon) through the incision through which the piece is obtained, and the anastomosis is performed. It does not require, therefore, an important training in intracorporeal sutures. On the contrary, it forces to make the abdominal incision in the area that allows the extraction of said ends. In obese patients it can be difficult since the mesos are short and do not allow their extraction easilywith ,so sometimes, it forces excessive traction. In addition, intestinal rotations during the anastomosis may go unnoticed.

Although there are currently defenders of both techniques, the extracorporeal anastomosis is currently the most performed in our environment and will be used as a reference treatment in the present study.

Numerous studies have been published comparing both techniques. A very recent meta-analysis, including 12 non-randomized comparative studies with 1492 patients, concluded that intracorporeal anastomosis is associated with less morbidity and a reduction in hospital stay, suggesting a faster recovery. To date, no well-designed, prospective, randomized and randomized study exists in the literature. We believe it is necessary, therefore, to carry out a project that compares both surgical techniques in the treatment of right colon cancer and assess which is associated with a lower postoperative morbidity.

ELIGIBILITY:
Inclusion Criteria:

* All patients had to be 18 years of age or over, to be programmed for laparoscopic surgery for right colon neoplasm and provide a signed written consent form.

Exclusion Criteria:

* All patients who do not meet all the inclusion criteria were excluded. The other exclusion criteria included the need for emergency surgery, renal failure defined by haemodialysis, Crohn's disease, ulcerative colitis, T4 tumor invading adjacent organs, synchronous colorectal neoplasm, metastasis or carcinomatosis at diagnosis, bowel obstruction, psychiatric disorders or contraindication for laparoscopic approach.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
In patients with right colon cancer, laparoscopic right hemicolectomy with intracorporeal anastomosis presents less perioperative morbidity than extracorporeal anastomosis. | 24 months
  To compare perioperative morbidity between laparoscopic right hemicolectomy with intracorporeal anastomosis versus extracorporeal anastomosis within 30 days after surgery.

SECONDARY OUTCOMES:
Surgical time | 4 hours
  o evaluate the difference in surgical time between right hemicolectomy with intracorporeal versus extracorporeal anastomosis.
VAS | 24 hour
  Quantify, by means of the Visual-Analogue Scale (VAS: is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity. Based on the distribution of pain VAS scores in post- surgical patients who described their postoperative pain intensity as none, mild, moderate, or severe, the following cut points on the pain VAS have been recommended: no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm)), postoperative pain 24 hours after surgery and the day of hospital discharge, and determine which of the two laparoscopic right hemicolectomy techniques produces less pain.
Dehiscence | 30 days
  To evaluate and compare the rate of anastomotic dehiscence in both groups of anastomoses up to 30 days after surgery.
Infection rate | 30 days
  To evaluate the infection rate of the surgical site in both groups up to 30 days after surgery.
Days of hospital stay | 180 days
  o compare the difference of days of hospital stay in both groups of anastomoses.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Ferrer-Marquez, Principal Investigator — Colorectal Surgeon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jemal A, Siegel R, Ward E, Hao Y, Xu J, Thun MJ. Cancer statistics, 2009. CA Cancer J Clin. 2009 Jul-Aug;59(4):225-49. doi: 10.3322/caac.20006. Epub 2009 May 27. PMID 19474385
- [Background] Bilimoria KY, Palis B, Stewart AK, Bentrem DJ, Freel AC, Sigurdson ER, Talamonti MS, Ko CY. Impact of tumor location on nodal evaluation for colon cancer. Dis Colon Rectum. 2008 Feb;51(2):154-61. doi: 10.1007/s10350-007-9114-2. Epub 2008 Jan 3. PMID 18172729
- [Background] Le Voyer TE, Sigurdson ER, Hanlon AL, Mayer RJ, Macdonald JS, Catalano PJ, Haller DG. Colon cancer survival is associated with increasing number of lymph nodes analyzed: a secondary survey of intergroup trial INT-0089. J Clin Oncol. 2003 Aug 1;21(15):2912-9. doi: 10.1200/JCO.2003.05.062. PMID 12885809
- [Background] Jacobs M, Verdeja JC, Goldstein HS. Minimally invasive colon resection (laparoscopic colectomy). Surg Laparosc Endosc. 1991 Sep;1(3):144-50. PMID 1688289
- [Background] Colon Cancer Laparoscopic or Open Resection Study Group; Buunen M, Veldkamp R, Hop WC, Kuhry E, Jeekel J, Haglind E, Pahlman L, Cuesta MA, Msika S, Morino M, Lacy A, Bonjer HJ. Survival after laparoscopic surgery versus open surgery for colon cancer: long-term outcome of a randomised clinical trial. Lancet Oncol. 2009 Jan;10(1):44-52. doi: 10.1016/S1470-2045(08)70310-3. Epub 2008 Dec 13. PMID 19071061
- [Background] Hazebroek EJ; Color Study Group. COLOR: a randomized clinical trial comparing laparoscopic and open resection for colon cancer. Surg Endosc. 2002 Jun;16(6):949-53. doi: 10.1007/s00464-001-8165-z. Epub 2002 Mar 18. PMID 12163961
- [Background] Jayne DG, Guillou PJ, Thorpe H, Quirke P, Copeland J, Smith AM, Heath RM, Brown JM; UK MRC CLASICC Trial Group. Randomized trial of laparoscopic-assisted resection of colorectal carcinoma: 3-year results of the UK MRC CLASICC Trial Group. J Clin Oncol. 2007 Jul 20;25(21):3061-8. doi: 10.1200/JCO.2006.09.7758. PMID 17634484
- [Background] Lacy AM, Garcia-Valdecasas JC, Delgado S, Castells A, Taura P, Pique JM, Visa J. Laparoscopy-assisted colectomy versus open colectomy for treatment of non-metastatic colon cancer: a randomised trial. Lancet. 2002 Jun 29;359(9325):2224-9. doi: 10.1016/S0140-6736(02)09290-5. PMID 12103285
- [Background] Kennedy GD, Heise C, Rajamanickam V, Harms B, Foley EF. Laparoscopy decreases postoperative complication rates after abdominal colectomy: results from the national surgical quality improvement program. Ann Surg. 2009 Apr;249(4):596-601. doi: 10.1097/SLA.0b013e31819ec903. PMID 19300230
- [Background] Wu Q, Jin C, Hu T, Wei M, Wang Z. Intracorporeal Versus Extracorporeal Anastomosis in Laparoscopic Right Colectomy: A Systematic Review and Meta-Analysis. J Laparoendosc Adv Surg Tech A. 2017 Apr;27(4):348-357. doi: 10.1089/lap.2016.0485. Epub 2016 Oct 21. PMID 27768552
- [Background] Milone M, Elmore U, Di Salvo E, Delrio P, Bucci L, Ferulano GP, Napolitano C, Angiolini MR, Bracale U, Clemente M, D'ambra M, Luglio G, Musella M, Pace U, Rosati R, Milone F. Intracorporeal versus extracorporeal anastomosis. Results from a multicentre comparative study on 512 right-sided colorectal cancers. Surg Endosc. 2015 Aug;29(8):2314-20. doi: 10.1007/s00464-014-3950-7. Epub 2014 Nov 21. PMID 25414066
- [Background] Ricci C, Casadei R, Alagna V, Zani E, Taffurelli G, Pacilio CA, Minni F. A critical and comprehensive systematic review and meta-analysis of studies comparing intracorporeal and extracorporeal anastomosis in laparoscopic right hemicolectomy. Langenbecks Arch Surg. 2017 May;402(3):417-427. doi: 10.1007/s00423-016-1509-x. Epub 2016 Sep 5. PMID 27595589
- [Background] Shapiro R, Keler U, Segev L, Sarna S, Hatib K, Hazzan D. Laparoscopic right hemicolectomy with intracorporeal anastomosis: short- and long-term benefits in comparison with extracorporeal anastomosis. Surg Endosc. 2016 Sep;30(9):3823-9. doi: 10.1007/s00464-015-4684-x. Epub 2015 Dec 10. PMID 26659237
- [Background] Carnuccio P, Jimeno J, Pares D. Laparoscopic right colectomy: a systematic review and meta-analysis of observational studies comparing two types of anastomosis. Tech Coloproctol. 2014 Jan;18(1):5-12. doi: 10.1007/s10151-013-1029-4. Epub 2013 May 18. PMID 23686680
- [Background] Morpurgo E, Contardo T, Molaro R, Zerbinati A, Orsini C, D'Annibale A. Robotic-assisted intracorporeal anastomosis versus extracorporeal anastomosis in laparoscopic right hemicolectomy for cancer: a case control study. J Laparoendosc Adv Surg Tech A. 2013 May;23(5):414-7. doi: 10.1089/lap.2012.0404. PMID 23627922
- [Background] Feroci F, Lenzi E, Garzi A, Vannucchi A, Cantafio S, Scatizzi M. Intracorporeal versus extracorporeal anastomosis after laparoscopic right hemicolectomy for cancer: a systematic review and meta-analysis. Int J Colorectal Dis. 2013 Sep;28(9):1177-86. doi: 10.1007/s00384-013-1651-7. Epub 2013 Feb 1. PMID 23371336
- [Background] Lee KH, Ho J, Akmal Y, Nelson R, Pigazzi A. Short- and long-term outcomes of intracorporeal versus extracorporeal ileocolic anastomosis in laparoscopic right hemicolectomy for colon cancer. Surg Endosc. 2013 Jun;27(6):1986-90. doi: 10.1007/s00464-012-2698-1. Epub 2013 Jan 9. PMID 23299132
- [Background] Cirocchi R, Trastulli S, Farinella E, Guarino S, Desiderio J, Boselli C, Parisi A, Noya G, Slim K. Intracorporeal versus extracorporeal anastomosis during laparoscopic right hemicolectomy - systematic review and meta-analysis. Surg Oncol. 2013 Mar;22(1):1-13. doi: 10.1016/j.suronc.2012.09.002. Epub 2012 Oct 30. PMID 23116767
- [Background] van Oostendorp S, Elfrink A, Borstlap W, Schoonmade L, Sietses C, Meijerink J, Tuynman J. Intracorporeal versus extracorporeal anastomosis in right hemicolectomy: a systematic review and meta-analysis. Surg Endosc. 2017 Jan;31(1):64-77. doi: 10.1007/s00464-016-4982-y. Epub 2016 Jun 10. PMID 27287905
- [Result] Wong JT, Abbas MA. Laparoscopic right hemicolectomy. Tech Coloproctol. 2013 Feb;17 Suppl 1:S3-9. doi: 10.1007/s10151-012-0931-5. Epub 2012 Dec 19. PMID 23250636
- Available data/document: Study Protocol: Proyect — https://drive.google.com/file/d/1EEFxi3XpaRW12IAzVctIrrOSo6EKi70_/view?usp=sharing — A project that compares both surgical techniques in the treatment of right colon cancer and assess which is associated with a lower postoperative morbidity

DOCUMENTS (1):
  • Study Protocol (2016-01-01): https://cdn.clinicaltrials.gov/large-docs/14/NCT03990714/Prot_000.pdf